CLINICAL TRIAL: NCT00335231
Title: The Effect of Preoperative Topical Gatifloxacin on Anterior Chamber Sample Cultures After Cataract Surgery.
Brief Title: Preoperative Topical Gatifloxacin on Anterior Chamber Cultures After Cataract Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol changes underway. Trial never started
Sponsor: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QUEENS-SRE-3
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Endophthalmitis
Keywords: Post-cataract surgery endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Gatifloxacin

ARMS (2):
- gatifloxacin (Experimental): one group will receive topical application of gatifloxacin prior to surgery,
  Interventions: Drug: gatifloxacin ophthalmic (ZYMAR)
- no eye drops (No Intervention): this group will receive no eye drops.

INTERVENTIONS:
Drug: gatifloxacin ophthalmic (ZYMAR)
  Arms: gatifloxacin

SUMMARY:
Postoperative endophthalmitis, a possible severe complication of cataract surgery, is an infection of the anterior chamber of the eye caused by bacterial contamination and colonization through surgical incisions. Bacteria are thought to originate mainly from the patient's skin and studies show that bacteria are commonly found in the anterior chamber following surgery. However, innate immune defences are usually able to control and eliminate bacterial growth before postoperative endophthalmitis occurs. Also, due to the low incidence of postoperative endophthalmitis, it is difficult to accurately evaluate preventative methods. This study will examine the efficacy of topical preoperative administration of gatifloxacin (a new fourth generation fluoroquinolone antibiotic) on reduction of bacterial contamination of the anterior chamber following cataract surgery. If the antibiotic is shown to lower bacteria count in cultures from anterior chamber fluid, it has the potential to lower the incidence of postoperative endophthalmitis.

Patients undergoing cataract surgery will be notified and asked to participate in the study by the physician in advance of the surgery, provided they do not possess any exclusion criteria. The participants will be randomly split into two groups; one group will receive topical application of gatifloxacin prior to surgery, while the other group will receive no eye drops. During surgery, a small sample of anterior chamber fluid will be removed from the eye and cultured in both broth and enrichment media for all subjects. Bacterial growth, i.e., colony forming units (CFUs), will be used as an indicator of the bacterial contamination of the fluid.

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery on first eye (i.e., first cataract surgery.

Exclusion Criteria:

* uveitis,
* herpetic eye disease,
* corneal ulceration,
* severe blepharitis,
* past trauma to the eye,
* complicated cataract surgery (e.g., posterior capsule rupture),
* previous intraocular surgeries.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Difference in bacterial colony forming units (CFUs) between treatment (gatifloxacin) and no treatment group

SECONDARY OUTCOMES:
Bacterial sensitivity
Patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Defrawy, MD PhD FRCSC, Principal Investigator — Queen's University, Hotel Dieu Hospital, Kingston General Hospital
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada